CLINICAL TRIAL: NCT04298047
Title: A 3-month Cycle of Weekly Montreal Museum of Fine Arts Tours to Promote Social Inclusion, Well-being, Quality of Life and Health in Older Community Members Experiencing Social Isolation
Brief Title: A 3-month Cycle of Weekly Montreal Museum of Fine Arts Tours
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, PhD, Professor of Geriatrics, Holder of the Dr. Joseph Kaufmann Chair in Geriatric Medicine Clinician Scientist, Department of Medicine, Division of Geriatric Medicine Director of Centre of Excellence on Longevity, RUISSS McGill, McGill University, Jewish General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 20201789
Record Dates: First submitted 2020-03-04; First posted 2020-03-06 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Social Interaction; Quality of Life; Health
Keywords: Community-dwellers; older adults; museum; art

STUDY DESIGN:
Intervention Model Description: The design is a unicentre (Jewish General Hospital; Montreal, Quebec, Canada), clinical, randomized, controlled, single blinded (i.e.; investigators), superiority trial, with two parallel arms (Intervention and Control groups), comparative (comparison between Intervention and Control groups) and analyzed with the intention-to-treat.
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): The participants in the Intervention group will be participants of the MMFA participatory art-based activity.
  Interventions: Other: participatory art-based activity
- Control Group (No Intervention): The Control arm will be composed of older community dwellers matched on age and sex compared to the Intervention group but who will not be participants at the MMFA participatory art-based activity.

INTERVENTIONS:
Other: participatory art-based activity — The intervention is a 3-month cycle of weekly guided tours carried out at the MMFA. Each visit will be performed with a group of 8 participants and a trained guide. They will meet at the museum once per week for a 45 min museum guided tour during a 3-month period. Each visit will be different and supervised by a museum guide. Regardless the topic of the visits, each visit will be standardized and separated in two consecutive phases: (1) Presentation of the objectives of the activity and (2) tour with a guide. Guided tours will target visual art (i.e., painting). They will be tailor-made and based on emotions and interactions in front of painting. The levels of information given to participants will regularly (i.e., each month) increase during the 3-month cycle of museum guided tours. The participants will be separated in 8 groups of 8 individuals per week. The same guide will manage each group of 8 participants during the 12 planned visits.
  Arms: Intervention group

SUMMARY:
Social isolation in older community-members living in urban areas and its possible reduction through a 3-month cycle of weekly museum tours.

DETAILED DESCRIPTION:
Social isolation is a major problem for the Canadian society because of its: (1) high prevalence in the older population (30% in individuals aged 65 and over, which represents 1.5 million individuals), (2) association with a wide range of mental and physical health problems and (3) increased use of health and social services. Museum art-based activities have demonstrated benefits on an individual's sense of social inclusion, their well-being, their quality of life and physical frailty. Few studies have examined the effects of the participation in museum art-based activities in older community members experiencing social isolation. In 2019, the team conducted an experimental pilot study comprised of pre-post intervention, single arm, prospective and a longitudinal follow-up. This experiment indicated that a 3-month cycle of weekly visits to the Montreal Museum of Fine Arts (MMFA) in the form of a guided tour may improve the social inclusion of socially isolated older adults. We hypothesize that it is possible to reproduce these previous positive results using a mixed methods approach that combines: (1) a qualitative phase comprised of observation of the guided tours; semi-structured interviews, focus groups and an analysis of relevant organizational documents; (2) a quantitative phase based on a randomized clinical trial (RCT). Over a two-year period, we will examine whether and how a 3-month cycle of weekly MMFA tours may (1) improve social inclusion, well-being and quality of life, and (2) reduce frailty in older community members, living in Montreal, who are experiencing social isolation. The study includes the participation of community workers who work with socially isolated older Montrealers, members of this community, as well as museum works and administrators. Our research will not only include information on how the museum experience has affected older adults. It will incorporate feedback from all of these participants leading to an evaluation of the program offered by the museum to better serve the future needs and desires of this population. It will also benefit the participating organizations.

ELIGIBILITY:
Inclusion Criteria:

1. Being 65 years and over
2. Having an Internet access with an electronic device (i.e.; laptop, computer, smartphone, tablet) at the participant's place of living as the repetitive assessments for this study will be performed on the web platform of the Centre of Excellence on Longevity of McGill University
3. Understanding and writing the language of the recruitment centre (i.e., French or English)
4. Life expectancy estimated over 3 months as the duration of the follow-up is 3 months

Exclusion Criteria:

1. Concomitant participation to another clinical trial,
2. Having participated to a participatory art-based activity of the MMFA,
3. Not speaking the language of the study.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Social isolation | 3 months
  The 11-item Duke Social Support Index (DSSI) comprises two subscales: social interaction (i.e., frequency of interactions) and subjective support (i.e., satisfaction with emotional support provided). DSSI score ranges from 11 to 33, increased score indicating higher levels of social insertion. The scores of the 11 items are combined and categorized as low-fair (score ≤26), high (score 27-29) and very high (score 30-33). We will use as primary outcome the mean score of 11-item DSSI and its distribution in three categories.

SECONDARY OUTCOMES:
Frailty | 3 months
  The Centre of Excellence on longevity Self-AdMinistered questionnaire (CESAM). This questionnaire is composed of 20 items examining different domains including weight loss; polypharmacy; vision, hearing and memory issues; use of home support (i.e., family, friend and/or professional); the activity of daily living and the instrumental activity daily living scales; mood; practice of regular physical activity and history of falls in the past 12 months.
Well-being | 3 months
  Assessed using the Warwick-Edinburgh Mental Well-being Scale (WEMWBS) questionnaire. The WEMWBS covers most aspects of positive mental health (positive thoughts and feelings). Its score ranges from 14 (i.e., none of the time) to 70 (i.e., all the time)
Quality of life using the EuroQol-5D (EQ-5D) | 3 months
  EuroQol-5D self-questionnaire, evaluating mobility, usual activities, self-care, pain, anxiety and mood, from No problem to Unable, scored from 5 to 25, High score meaning a bad quality of life.
Participants' socio-demographic characteristics | 3 months
  i.e., age, sex, marital status defined as married, living common-law, single, separated, divorced or widowed, place of living defined as home versus residence) and low household income using Canadian low-income cut-off
Interpersonal interactions | 3 months
  evaluation adapted from Observed Emotions Rating Scale (OERS). The OERS is about the completion of observations of 5 categories listed in order to give an overall look at the participants' interpersonal interactions based on expression of emotions. The 5 categories are; 1/ pleasure, 2/ anger, 3/ anxiety/fear, 4/ sadness, 5/ general alertness.
Compliance assessed counting the number of workshops completed during the 3-month period of intervention. | 3 month
  assessed counting the number of workshops completed during the 3-months period of intervention.
Satisfaction concerning the project assessed by self-questionnaire | 1 day
  self-questionnaire, qualitative (from 1 to 10: Dissatisfying to Satisfying), NO GLOBAL SCORE, each question is evaluated separately. A mean of all questions to have a global note (/10) will eventually be done for each participant.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — McGill University
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No